CLINICAL TRIAL: NCT04989387
Title: A Phase 1, Open-Label, Multicenter Study of INCA00186 as Monotherapy or in Combination With Immunotherapy in Participants With Advanced Solid Tumors
Brief Title: Study of INCA 0186 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was a strategic business decision. There were no safety concerns contributing to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: INCA 0186-101; 2021-001263-24 (EudraCT Number)
Record Dates: First submitted 2021-07-22; First posted 2021-08-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors; Squamous Cell Carcinoma of the Head and Neck (SCCHN); Gastrointestinal (GI) Malignancies
Keywords: open label; advanced solid tumors; squamous cell carcinoma of the head and neck; gastrointestinal malignancies; gastric/gastroesophageal junction cancer; hepatocellular carcinoma; pancreatic ductal adenocarcinoma; squamous carcinoma of the anal canal; colorectal cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Group A Dose Escalation and Expansion (Experimental): INCA00186 will be administered as monotherapy every 2 or every 4 weeks.
  Interventions: Drug: INCA00186
- Treatment Group B1 Dose Escalation and Expansion (Experimental): INCA00186 will be administered in combination with retifanlimab. INCA00186 will be administered every 2 or 4 weeks and retifanlimab will be administered every 4 weeks.
  Interventions: Drug: INCA00186; Drug: Retifanlimab
- Treatment Group B2 Dose Escalation and Expansion (Experimental): INCA00186 will be administered in combination with INCB106385. INCA00186 will be administered every 2 or 4 weeks and INCB106385 will be administered once or twice daily.
  Interventions: Drug: INCA00186; Drug: INCB106385
- Treatment Group C Dose Escalation and Expansion (Experimental): INCA00186 will be administered in combination with retifanlimab and INCB106385. INCA00186 will be administered every 2 to 4 weeks, retifanlimab every 4 weeks and INCB106385 once or twice daily.
  Interventions: Drug: INCA00186; Drug: Retifanlimab; Drug: INCB106385

INTERVENTIONS:
Drug: INCA00186 — INCA00186 will be administered every 2 weeks or 4 weeks as per protocol
Drug: Retifanlimab — Retifanlimab will be administered every 4 weeks as per protocol
  Arms: Treatment Group B1 Dose Escalation and Expansion; Treatment Group C Dose Escalation and Expansion
Drug: INCB106385 — INCB106385 will be administered orally once or twice a day.
  Arms: Treatment Group B2 Dose Escalation and Expansion; Treatment Group C Dose Escalation and Expansion

SUMMARY:
This is an open-label, nonrandomized, multicenter, dose escalation, and dose expansion first-in human (FIH) Phase 1 study to determine the safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of INCA00186 when given alone or in combination with INCB106385 and/or retifanlimab in participants with specific advanced solid tumors; squamous cell carcinoma of the head and neck (SCCHN) and specified gastrointestinal (GI) malignancies have been selected as indications of interest for this study. Participants with CD8 T-cell-positive tumors will be selected as these tumors are more likely to respond to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Male or female participant aged 18 years or older inclusive at the time of signing the ICF.
* Must be willing and able to conform to and comply with all Protocol requirements
* Willingness to undergo pre- and on-treatment tumor biopsy.
* Have CD8 T-cell-positive tumors
* ECOG performance status 0 or 1.
* Measurable disease according to RECIST v1.1.
* Participants with SCCHN: Participants with histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx not amenable to local therapy with curative intent (surgery or radiation with or without chemotherapy).
* Participants with specified GI malignancies: Histologically or cytologically confirmed advanced or metastatic colorectal (CRC), gastric/gastroesophageal junction (GEJ) cancer, hepatocellular carcinoma (HCC), pancreatic ductal adenocarcinoma (PDAC), or squamous carcinoma of the anal canal (SCAC).
* Participants should have disease progression after treatment with available therapies, including anti-PD-(L)1 therapy (if applicable), that are known to confer clinical benefit or who are intolerant to or ineligible for standard treatment. Prior anti-PD-(L)1 therapy should not have been discontinued because of intolerance.
* For participants to be enrolled in cohorts including INCB106385: The ability to swallow oral medication.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Clinically significant cardiac disease, unstable angina, acute myocardial infarction within 6 months of Cycle 1 Day 1, and New York Heart Association Class III or IV congestive heart failure.
* History or presence of an ECG abnormality that, in the investigator's opinion, is clinically meaningful.
* Known active CNS metastases and/or carcinomatous meningitis.
* Participants who have active or inactive autoimmune disease or syndrome (eg, rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (doses > 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of the first dose of study treatment with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the participant has been disease free > 1 year after treatment with curative intent.
* Participants with protocol specified exclusionary hematology, hepatic, renal and coagulation laboratory values at screening.

Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting study treatment.

* Evidence of interstitial lung disease, history of interstitial lung disease, or active noninfectious pneumonitis.
* Immune-related toxicity during prior immune therapy for which permanent discontinuation of therapy is recommended, OR any immune-related toxicity requiring intensive or prolonged immunosuppression to manage.
* Prior treatment with any adenosine pathway targeting drugs.
* Any prior chemotherapy, biological therapy, or targeted therapy to treat the participant's disease within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* Any prior radiation therapy within 28 days before the first dose of study treatment.
* Undergoing treatment with another investigational medication or having been treated with an investigational medication within 5 half-lives or 28 days (whichever is shorter) before the first dose of study treatment.
* For participants to be enrolled in cohorts including INCB106385: concomitant treatment with strong CYP3A4 inhibitors or inducers.
* Receipt of a live virus vaccine within 30 days of the first dose of study treatment.
* Infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week of the first dose of study treatment.
* Known or suspected SARS-CoV-2 infection at the time of enrollment.
* Active HBV or HCV infection that requires treatment. HBV-DNA and HCV-RNA must be undetectable. Participants who have cleared a prior HBV infection (defined as HBsAg negative, HBsAg antibody positive, and anti-HBc antibody positive) are eligible for the study.
* Known history of HIV (HIV 1/2 antibodies).
* History of organ transplant, including allogeneic stem-cell transplantation or CAR-T cell therapy.
* Known hypersensitivity or severe reaction to any component of study drug(s) or formulation components.
* For participants to be enrolled in cohorts including INCB106385: Inability to swallow food or any concomitant condition of the upper GI tract that precludes administration of oral medications.
* Is pregnant or breastfeeding.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* The following participants are excluded in France: vulnerable populations according to article L.1121-6 of the French Public Health Code and adults under legal protection or who are unable to express their consent per article L.1121-8 of the French Public Health Code.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of INCA00186 as monotherapy and in combination with retifanlimab and/or INCB106385 as measured by the number of participants with adverse eventsductions and withdrawal of treatment due to AEs | 90 days after study completion totaling up to 27 months
Evaluation of Dose-Limiting Toxicity (DLTs) of INCA00186 as monotherapy and in combination with retifanlimab and/or INCB106385 as measured by safety events during treatment | 90 days after study completion totaling up to 27 months
Evaluation of Recommended Dose for Expansion (RDE) of INCA00186 as monotherapy and in combination with retifanlimab and/or INCB106385 as measured by safety, PK and PD data | 90 days after study completion totaling up to 27 months

SECONDARY OUTCOMES:
Determination of PK parameter Maximum Observed Plasma Concentration (Cmax) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Determination of PK parameter of Time to Maximum Plasma Concentration (tmax) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Determination of PK parameter of concentration at the end of the dosing interval (Ctau) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Determination of PK parameter of area under the plasma or serum concentration-time curve (AUC) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Determination of PK parameter of total clearance (CL) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Determination of PK parameter of volume of distribution (Vz) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Determination of PK parameter half-life (t1/2) for INCA00186 | Cycle 1 days 1, 2, 8, 15, 22; Cycle 2 days 1, 8; Day 1 of every other cycle starting at Cycle 4 (ie, Cycle 4 day 1, Cycle 6 day 1, etc; each cycle is 28 days) + 30 day follow-up; approximately 24 months
Intratumoral effect of INCA0186 on CD73 enzymatic activity | 2 biopsy samples will be taken: pre-treatment and on-treatment on Cycle 1 Day 22 (for every 2 week INCA00186 dosing group) or Cycle 2 Day 8 (for every 4 week INCA00186 dosing group); each cycle is 28 days; sampling will be taken within 2 months.
Objective Response Rate (ORR) by radiographic disease assessment | Baseline through end of study up, to 24 months
Disease Control Response (DCR) determined by radiographic disease assessment | Baseline through end of study, up to 24 months
Duration of Response (DOR) from earliest date of disease response until earliest date of disease progression as determined by radiographic disease assessment, or death if occurring sooner than progression | Baseline through end of study, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Rybicka, MD, Study Director — Incyte Corporation
Locations (32):
- United States (8):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Carolina Bio-Oncology Institute, Pllc, Huntersville, North Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Austria (2):
  - Innsbruck University Hospital, Innsbruck
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (5):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Ghent University Hospital, Ghent
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
- Netherlands (5):
  - Netherlands Cancer Institute Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud University Nijmegen Medical Center, Nijmegen
  - Erasmus Mc Cancer Institute, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Spain (6):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Institut Catala Doncologia Ico - Hospital Duran I Reynals Location, Barcelona
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
- United Kingdom (6):
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Guys and St Thomas Nhs Foundation Trust, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - Freeman Hospital Newcastle Upon Tyne Foundation Nhs Trust, Newcastle upon Tyne
  - The Royal Marsden Nhs Foundation Trust - Chelsea, Sutton

IPD SHARING:
Plan to Share IPD: No